CLINICAL TRIAL: NCT07191366
Title: EXPRESSMOM2 in Pregnant Women at High Risk of Preterm Birth. Aspects of Antenatal Breastmilk Expression and Safety From Gestational Week 28-34 and Potential Nutritional Benefits for the Newborn Infant.
Brief Title: Antenatal Breastmilk Expression in Pregnant Women at High Risk of Preterm Birth
Acronym: EXPRESSMOM2
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Odense University Hospital (Other)
Collaborators: Aabenraa Hospital (Other); Esbjerg Hospital - University Hospital of Southern Denmark (Other); Kolding Sygehus (Other); University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: OUH-HCA042
Record Dates: First submitted 2025-09-01; First posted 2025-09-24 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-08

CONDITIONS: Preterm Birth; PPROM; Preeclampsia; Previous Preterm Birth
Keywords: Antenatal breastmilk expression; ABME; Preterm birth; PPROM; Preeclampsia; Previous preterm birth; Colostrum; Colostrum analysis; Safety; self-efficacy
MeSH Terms: conditions — Premature Birth; Preterm Premature Rupture of the Membranes; Pre-Eclampsia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Handstimulation of the breasts (Experimental): Antenatal breastmilk expression and colostrum collection
  Interventions: Procedure: Handstimulation of breast
- Control (No Intervention)

INTERVENTIONS:
Procedure: Handstimulation of breast — Hand stimulation of the breast
  Other Names: aBME; Breastmilk expression
  Arms: Handstimulation of the breasts

SUMMARY:
In this randomized controlled study, the investigators aim to examine if antenatal breastmilk expression (aBME) from week 28 in high-risk pregnancies is a safe and effective method to ensure early access to mother's own milk.

In addition, this study will analyze and compare colostrum from pregnancy with colostrum after birth, investigates women's confidence in breastfeeding and breastfeeding establishment as well as measures oxytocin levels during aBME and active labour with no aBME.

DETAILED DESCRIPTION:
In this study 250 pregnant women at high risk of preterm birth (Diagnosed with either preeclampsia or PPROM or previously delivered preterm before week 34) from the Region of Southern Denmark, will be randomized into an intervention or a control group.

Women in the intervention group will be instructed to perform antenatal breastmilk expression twice daily for 5 minutes on each breast from inclusion at week 28-34 until birth. Women will be advised to collect any expressed milk and bring to the delivery ward for use after birth.

A total of 40 minutes of Cardio Toco Graphy (CTG) will be performed before, during and after they perform aBME for the first time, to detect any uterine contractions or foetal compromise due to stimulation. If the CTG is normal the women can begin aBME at home.

Furthermore, the women will be asked to answer a questionnaire about breastfeeding self-efficacy at inclusion and 2 weeks after aBME starts. Small amounts of the colostrum expressed before and after birth will be analysed for specific proteins, bioactive components and amount and types of Lactobacillus strains.

Women admitted to Odense University Hospital will be asked for a single blood sample to measure oxytocin. Samples will be drawn during the first aBME and at birth.

8 women/parents will be asked to participate in an observational study. Observations will follow breastfeeding practices within the first two days and afterward, weekly, during the first three weeks postpartum.

A subgroup of 12 mothers with a pre-pregnancy BMI above ≥30kg/m2 who give birth at term will be asked to participate in an in-depth face-to-face interview. The interviews will be conducted in the participant´s home 4-6 weeks postpartum to explore experiences with breastfeeding establishment after performing aBME.

The women in the control group will follow standard care and be asked to answer a questionnaire about breastfeeding self-efficacy at inclusion. Furthermore, women admitted to Odense University Hospital will be asked for a single blood sample to measure oxytocin. The sample will be drawn during randomization and at birth.

After birth, 8 women/parents will be asked to participate in an observational study. Observations will follow breastfeeding practices within the first two days and, afterward, weekly during the first three weeks.

The women from both groups will be followed until 6 months postpartum to monitor outcomes related to breastfeeding, nutrition, growth, and infections. Until four weeks after the infant's corrected age, all women in both groups receive weekly push messages through the smartphone application, including questions on feeding postpartum. If admitted, the feeding will be registered at the hospital through electronic health records. The following five months, all women in both groups will receive monthly push messages through the smartphone application, including post-partum feeding questions.

Furthermore, all women will be asked to answer a questionnaire related to breastfeeding self-efficacy 3 weeks after birth.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women with a GA between 28 weeks and 0 days and 34 weeks and 0 days who are either diagnosed with preeclampsia or PPROM or have previously given birth before 34 weeks of gestation
* Resident in the Region of Southern Denmark
* Women speaking and understanding Danish or English
* Planning to breastfeed their infants

Exclusion Criteria:

* HELLP or severe preeclampsia indicating expected induction of labour/caesarean section within a few days (According to national guidelines)
* Chorioamnionitis indicating induction of labour/caesarean section within a few days
* Women with a vaginal cerclage and PPROM
* Women taking medications contraindicating breastfeeding
* Women with prior breast reductive surgery or mastectomy
* Below 18 years of age
* Contractions to a certain extend expecting delivery within a few days
* Included in other trials, where breastfeeding is among outcomes

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2026-09 (Estimated); Primary Completion 2029-01 (Estimated); Study Completion 2029-07 (Estimated)

PRIMARY OUTCOMES:
Number of days from randomization to birth | From date of randomization at 28 weeks to 34 weeks of pregnancy until the date of birth. Up to 100 days.
  To investigate the safety of antenatal breastmilk expression in pregnant women at high risk of preterm birth included from week 28 to 34 of pregnancy

SECONDARY OUTCOMES:
Amount of available mothers own milk at birth | At birth
  Availability of mothers own milk for the newborn infant after antenatal breastmilk expression in pregnancy
Oxytocin levels | At two time points. Baseline at randomization for the control group and during the first time with handstimulation of the breast in the intervention group. Second time point in both groups: During active labour.
  To compare oxytocin levels from performing antenatal breastmilk expression or not
Colostrum analysis | From pregnancy to one week after birth
  To characterize macronutrients, microbial and bioactive composition in colostrum expressed before and after birth
Postnatal outcomes in infants (Height in cm, weight in kg, hospital treatments, admittance to NICU, duration of admittance, occurence of infections, nutrition, early feeding, hypoglyceamia) | From date of birth to six months post partum.
  To compare feeding intolerance, risk of infection and NEC in infants fed only mothers own milk compared to mothers own milk and/or donor human milk
Maternal breastfeeding self-efficacy changes in questionnaires. | From date of randomization to 3 weeks post-partum
  To investigate if antenatal breastmilk expression affects maternal breastfeeding self-efficacy.
Breastfeeding establishment after antental breastmilk expression in obese women | At 4-6 weeks post-partum
  To examine experiences with breastfeeding establishment in women with obesity performing antenatal breastmilk expression or not
Observations regarding number of tools/strategies from antenatal breastmilk expression | Within the first 3 weeks of post-partum
  Number of tools and strategies in breastfeeding establishment after performing antenatal breastmilk expression in pregnancy
Number of women exclusively breastfeeding. | From date of birth to 3 weeks post partum.
  To investigate if antenatal breastmilk expression affects rates of exclusive breastfeeding

CONTACTS AND LOCATIONS:
Overall Officials: Gitte Zachariassen, MD, phd, Study Chair — The Hans Christian Andersen Children's Hospital, Odense University Hospital; Christina A Vinter, MD, phd, Study Chair — The Department of Gynaecology and Obstetrics, Odense University Hospital; Leonora S Borum, MD, Principal Investigator — The Hans Christian Andersen Children's Hospital, Odense University Hospital; Sarah B Bentzen, Midwife, Principal Investigator — The Hans Christian Andersen Children's Hospital, Odense University Hospital

IPD SHARING:
Plan to Share IPD: No